CLINICAL TRIAL: NCT03781570
Title: Brain and Genetic Predictors of Individual Differences in Pain and Analgesia
Acronym: PAINGEN
Status: Completed | Type: Observational
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: QIMR Berghofer Medical Research Institute (Other)
Responsible Party: Principal Investigator, Tor Wager, Director, Cognitive and Affective Neuroscience Laboratory; Professor, Department of Psychology and Neuroscience and the Institute for Cognitive Science, University of Colorado, Boulder
Other Study IDs: Pain Genetics
Record Dates: First submitted 2018-12-14; First posted 2018-12-20 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect saliva samples during the fMRI scan day and genotype using the same facility (same laboratory, personnel, platform, and protocols), following standard GWAS quality control procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: All participants are administered Control and Placebo creams (two interventions), with thermal and mechanical painful stimuli delivered repeatedly after each intervention. The order of intervention testing is Control, Placebo, Placebo, Control in a fixed order. All interventions are completed within a single testing session.
  Interventions: Behavioral: Placebo Cream; Behavioral: Control Cream

INTERVENTIONS:
Behavioral: Placebo Cream — In the Placebo intervention, participants are given an inert cream with instructions that it is "Prodicaine, an effective pain-relieving drug". The cream is applied to two fingers on the left hand.
Behavioral: Control Cream — In the Control intervention, participants are given an inert cream with instructions that it is "a control cream with no effects" . The cream is applied to two fingers on the left hand.

SUMMARY:
The purpose of the study is to gain a better understanding of pain processing in the brain. Our understanding of how pain is processed in the brain is limited. We are testing for individual differences in pain perception and emotion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be registered in the Colorado Community Twin Sample (CTS).

Exclusion Criteria:

* Not being registered in the Colorado Community Twin Sample (CTS).
* Any MRI contraindications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The CTS includes 727 same-sex twin pairs between 26-38 years old (as of Spring 2017), originally derived from the Colorado Twin Registry, a population based registry, housed at the Institute for Behavioral Genetics (IBG) at the University of Colorado since 1984, with three previous waves of data collection (1997-2002, 2002-2008, and 2009-2014).
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor Wager, PHD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado, Boulder, Boulder, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Main: All participants completed all conditions, with no groups/arms.
Period: Overall Study
Arm/Group | Main
Started | 541
Completed | 492
Not Completed | 49
Not completed — Technical Issues (equipment failure) | 31
Not completed — Withdrawal by Subject | 7
Not completed — Physical Constraints | 11

BASELINE CHARACTERISTICS:
Population: 32 participants (out of 492) were excluded from analysis: The first 10 participants completed a different experimental design (with different stimuli timing, intensities and ratings), 20 participants were excluded because all their pain ratings were with reaction time over the allotted time for rating or too short to be deliberate, one participant was insensitive to pain (due to their profession), and one participant was excluded due to data loss.
Arm/Group | Main
Number analyzed (Participants) | 460
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 460
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.25 (2.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272
  Male | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 434
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 4
  White | 418
  More than one race | 18
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 460

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating Scores Made on a Visual Analog Scale (VAS)
Description: Self reported pain using a Visual Analogue Scale (VAS) ranging from 0-100 (with 0 representing "no pain at all" and 100 representing "most intense pain imaginable (in the context of the experiment)). Higher scores indicate more pain. 0 is the minimum value and 100 is the maximum value. This scale is used for both thermal and mechanical pain. Reported values reflect averages of VAS ratings for individual stimuli for each of thermal and mechanical pain.
Time Frame: Measured during pain tasks at a single 4 hour experimental session (within one month of screening completion).
Population: All participants completed both the placebo condition and the control condition. Participants completed both conditions and all analyses were completed within participants. Descriptions of arms and interventions are detailed in the Protocol Section.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Main
Number analyzed (Participants) | 460
Score on a scale
  Placebo thermal pain ratings | 0.136 (0.123)
  Control thermal pain ratings | 0.190 (0.141)
  Placebo mechanical pain ratings | 0.126 (0.174)
  Control mechanical pain ratings | 0.160 (0.178)
Statistical Analysis 1: Comparison: Main; Comparing placebo vs. control for thermal pain ratings with mixed effects models controlling for the stimulus intensity and the familial structure of the data; Test type: Superiority; p < 0.001, Mixed Models Analysis; Satterthwaite's method was used to estimate degrees of freedom for the mixed effects model; Mean Difference (Final Values) = -0.0544, 95% CI 2-sided [-0.0648 to -0.0441], Standard Error of Mean 0.00517

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each participant during their participation (i.e., from the beginning to the end of their in person session). Participants were instructed to report any unusual events happening shortly after the experiment.
Description: one 4-hour session
Arm/Group | Main
All-Cause Mortality (participants affected / at risk) | 0/541
Serious Adverse Events (participants affected / at risk) | 0/541
Other Adverse Events (participants affected / at risk) | 0/541

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT03781570/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03781570/SAP_001.pdf